CLINICAL TRIAL: NCT06317740
Title: Effect of Green Management Intervention on Nurse Manager Outcomes: A Randomized Controlled Trial
Brief Title: Green Management Intervention Program For Nurse Managers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matrouh University (Other)
Responsible Party: Principal Investigator, Nagah Abd El-Fattah Mohamed Aly, Assistant professor of Nursing administration, Matrouh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 0306369
Record Dates: First submitted 2024-02-24; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Intervention; Knowledge, Attitudes, Practice
Keywords: Green; Management; Nurse Managers; Outcomes; Randomization
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial using two-group pretest-posttest designs
Who Masked: Participant
Masking Description: The study was carried out as a randomized controlled trial using two-group pretest-posttest designs in which the intervention group received an intervention program, in contrast to the comparison group. The study design of the present work followed the CONSORT 2010statement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): The intervention group received an intervention program.
  Interventions: Other: green management intervention program
- Comparison group (Other): The comparison group did not receive an intervention program.
  Interventions: Other: green management intervention program

INTERVENTIONS:
Other: green management intervention program — The program activities focused on integrating green management concepts into both theory and practice learning

SUMMARY:
Green management is the organization-wide strategy that aims to integrate environmental sustainability development into organizational management procedures for maintaining safety and striving high quality of care. The study aimed to examine the effect of a randomized trial of a green management intervention program on nurse manager outcomes.

DETAILED DESCRIPTION:
Green management is the organization-wide strategy that aims to integrate environmental sustainability development into organizational management procedures for maintaining safety and striving for high-quality care. The study aimed to examine the effect of a randomized trial of a green management intervention program on nurse manager outcomes.

The study design was a randomized controlled trial using two-group pretest-posttest designs, according to Consort's 2010 statement. The study was conducted on 100 nurse managers in each intervention and comparison group at Alexandria University Hospitals. Data was collected from April 2023 to December 2023 using questionnaires of nurse managers' knowledge of green management and nurse manager outcomes. The researchers met the nurse managers to clarify the study objectives and reply to any questions and queries. The data were collected using self-administrated questionnaires related to the personal demographic characteristics of nurse managers, nurse managers' knowledge of green management and nurse manager outcomes. The data were collected during the implementation of the green management intervention program.

ELIGIBILITY:
Inclusion Criteria:

Nurse managers

* Work in General wards, and critical and intensive care units.
* Willing to participate in the study.
* Sign informed consent.
* Have at least one year of experience.

Exclusion Criteria:

Nurse Managers

* Unwilling to participate in the study.
* Did not sign an informed consent.
* Absent from multiple training sessions or incompletely filled out the questionnaires.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Questionnaire to measure nurse managers' knowledge | three months
  Knowledge of 200 nurse managers as assessed using a binary scale (0= No, 1= Yes). Change in nurse managers' knowledge level in three months.
Questionnaires to measure nurse manager outcomes | six months
  Nurse manager outcomes (green commitment, engagement, and citizenship behaviors, in addition to the practice of green health care activities) as assessed by a five- Likert scale (From 1= disagree strongly to 5= agree strongly). Change in nurse manager outcomes in six months.

CONTACTS AND LOCATIONS:
Overall Officials: Nagah Abd El-Fattah Mohamed Aly, Ph.D, Study Chair — Faculty of Nursing, Matrouh University, Egypt; Wael M. Lotfy, Ph.D, Study Director — Faculty of Nursing, Matrouh University, Egypt
Locations (1):
- Faculty of Nursing, Matrouh University, Marsá Maţrūḩ, Egypt

IPD SHARING:
Plan to Share IPD: No